CLINICAL TRIAL: NCT00870610
Title: Cerebral Metabolism During Therapeutic Hypothermia for Cardiac Arrest
Brief Title: Jugular Venous Oxygen Saturation During Therapeutic Hypothermia After Cardiac Arrest
Acronym: SjO2
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: 2010
Record Dates: First submitted 2009-03-10; First posted 2009-03-27 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Hypoxic Brain Injury; Hypothermia
Keywords: jugular venous oxygen saturation; hypothermia
MeSH Terms: conditions — Hypoxia, Brain; Hypothermia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: retrograde jugular venous cannulation — Retrograde cannulation of jugular vein and intermittent sampling of venous blood from cerebral circulation before, during and after hypothermia.
  Other Names: SjO2, cerebrovenous oxygen saturation

SUMMARY:
The purpose of this study is to understand what happens to cerebral metabolism during therapeutic hypothermia for hypoxic brain injury following cardiac arrest.

DETAILED DESCRIPTION:
Latest international guidelines recommend the use of therapeutic hypothermia in patients who have had cardiac arrest and remain in coma after return of spontaneous circulation. This is recommended essentially to limit the cerebral injury caused by cardiac arrest and possibly amplified upon reperfusion. At times, although a spontaneous circulation has returned, cerebral oxygenation may remain inadequate due to inadequate perfusion pressure, and hypothermia, by reducing cardiac output and cerebral blood flow could actually aggravate this phenomenon. The rewarming period is thought to be at greatest risk of inadequate oxygenation for the increase in metabolic demand. With this study we aim to understand what happens to cerebral oxygenation and metabolism during therapeutic hypothermia for cardiac arrest through cerebrovenous oxygen saturation monitoring and in particular, to see whether through this type of monitoring we could recognize otherwise unnoticed periods of inadequate cerebral oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients in coma after cardiac arrest undergoing therapeutic hypothermia

Exclusion Criteria:

* Age < 18
* Pregnancy
* Traumatic brain injury
* Contraindications to cannulation as severe coagulopathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are in coma after cardiac arrest, admitted to the Intensive Care Unit of a University Teaching Hospital and undergoing therapeutic hypothermia
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Fondazione Ospedale Maggiore Policlinico Mangiagalli Regina Elena
Locations (1):
- Intensive Care Unit-Fondazione Ospedale Maggiore Policlinico Mangiagalli Regina Elena, Milan, Italy

REFERENCES:
- [Background] Nolan JP, Morley PT, Vanden Hoek TL, Hickey RW, Kloeck WG, Billi J, Bottiger BW, Morley PT, Nolan JP, Okada K, Reyes C, Shuster M, Steen PA, Weil MH, Wenzel V, Hickey RW, Carli P, Vanden Hoek TL, Atkins D; International Liaison Committee on Resuscitation. Therapeutic hypothermia after cardiac arrest: an advisory statement by the advanced life support task force of the International Liaison Committee on Resuscitation. Circulation. 2003 Jul 8;108(1):118-21. doi: 10.1161/01.CIR.0000079019.02601.90. No abstract available. PMID 12847056
- [Background] Bernard SA, Gray TW, Buist MD, Jones BM, Silvester W, Gutteridge G, Smith K. Treatment of comatose survivors of out-of-hospital cardiac arrest with induced hypothermia. N Engl J Med. 2002 Feb 21;346(8):557-63. doi: 10.1056/NEJMoa003289. PMID 11856794
- [Background] Macmillan CS, Andrews PJ. Cerebrovenous oxygen saturation monitoring: practical considerations and clinical relevance. Intensive Care Med. 2000 Aug;26(8):1028-36. doi: 10.1007/s001340051315. PMID 11030158